CLINICAL TRIAL: NCT06525077
Title: A Double-blind, Placebo-controlled, Randomized Withdrawal, Multicenter Study of the Efficacy and Safety of FT218 in the Treatment of Idiopathic Hypersomnia (IH)
Brief Title: Safety and Efficacy of FT218 in Idiopathic Hypersomnia (REVITALYZ)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Avadel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLFT218-2401
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-10

CONDITIONS: Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For the double-blind, randomized withdrawal portion of the study, the subject and all members of the study team will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FT218 (Experimental): FT218 at stable dose (selected during earlier titration) administered orally once nightly
  Interventions: Drug: FT218
- Placebo (Placebo Comparator): Placebo equivalent administered orally once nightly
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: FT218 — Sodium oxybate for extended-release oral suspension
  Other Names: LUMRYZ
  Arms: FT218
Other: Placebo — Matched placebo equivalent for oral suspension
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, randomized withdrawal, multicenter study of the efficacy and safety of FT218. FT218 drug product is a once-nightly formulation of sodium oxybate for extended-release oral suspension. The study will enroll subjects who are diagnosed with idiopathic hypersomnia. Subjects will be eligible to enroll regardless of current treatment with oxybate therapy or stimulants/alerting agents at study entry. The estimated total duration of study for each subject is approximately 18 weeks, including the Screening period.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of idiopathic hypersomnia
* Total ESS score at Screening > 11 if not on prior oxybate
* Average nightly total sleep time of > 7 hours
* May use stimulants/alerting agents but dose and regimen must have been stable for 2 months prior to Screening, and remain stable until the double-blind, randomized withdrawal visit
* Females of childbearing potential must use highly effective contraception for 2 months prior to Baseline, throughout the study, and for 30 days after the last dose of study drug
* Males with female partners of childbearing potential must use condoms throughout the study and for 30 days after the last dose of study drug
* Willing and able to provide informed consent and comply with the requirements of the study

Exclusion Criteria:

* Pregnant, nursing or lactating females
* Hypersomnia due to another medical, behavioral, sleep, or psychiatric condition
* Untreated or incompletely treated sleep apnea in patients with an apnea-hypopnea index (AHI) ≥ 15 by American Academy of Sleep Medicine (AASM) 1A criteria
* Clinically significant parasomnias
* History or presence of seizures, head trauma, succinic semialdehyde dehydrogenase deficiency, uncontrolled hypothyroidism, and/or significant hepatic impairment
* History or presence of bipolar and related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders
* Ongoing or past (within 1 year) major depressive episode
* At risk for suicide or history of suicide attempt
* If not on oxybate at Screening, treatment or planned treatment with any central nervous system (CNS) sedating agents during study
* Current or past substance use disorder (including alcohol or cannabinoids)
* Excessive caffeine consumption (> 600 mg/day)
* Prior treatment with either FT218 or LUMRYZ

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | End of stable dose visit to end of double-blind, randomized withdrawal visit [Week 12 to Week 14; 2 week period]
  Change in total ESS score

SECONDARY OUTCOMES:
Patient Global Impression of change (PGI-C) | End of stable dose visit to end of double-blind, randomized withdrawal visit [Week 12 to Week 14; 2 week period]
  Worsening of idiopathic hypersomnia symptoms as assessed by subject
Idiopathic Hypersomnia Severity Scale (IHSS) | End of stable dose visit to end of double-blind, randomized withdrawal visit [Week 12 to Week 14; 2 week period]
  Change in total IHSS score
Clinical Global Impression of change (CGI-C) | End of stable dose visit to end of double-blind, randomized withdrawal visit [Week 12 to Week 14; 2 week period]
  Worsening of idiopathic hypersomnia symptoms as assessed by clinician
Functional Outcomes of Sleep Questionnaire (FOSQ-10) | End of stable dose visit to end of double-blind, randomized withdrawal visit [Week 12 to Week 14; 2 week period]
  Change in total FOSQ-10 score

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Alpine Clinical Research Center, Boulder, Colorado
  - Florida Pediatric Institute, Winter Park, Florida
  - Clinical Research Institute, Stockbridge, Georgia
  - Clinical Neurophysiology Services PC, Sterling Heights, Michigan
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Tidewater Physicians Multispecialty Group (TPMG) Clinical Research, Williamsburg, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: REVITALYZ Study Website — http://www.revitalyz.com